CLINICAL TRIAL: NCT05346016
Title: Multigenerational Gut Bacteria Transmission and Its Stability in Families
Brief Title: The PEARL-AGE Study. Multigenerational Gut Bacteria Transmission and Its Stability in Families.
Status: Enrolling by invitation | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Earlham Institute (Unknown); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Other Study IDs: QIB01-2021
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Family Research
Keywords: gut microbiome; microbial adaptation; microbial evolution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples will be collected from the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators will recruit up to 4-generations of human family cohorts, in order to characterize the microbiome and its changes across different generations.

DETAILED DESCRIPTION:
Interest in the gut microbiome from both the scientific community and public has increased exponentially over the last decade. Yet our knowledge of the microbes in the gut microbiome, their persistence and dispersal to new human hosts is still surprisingly ill-defined.

Investigators hypothesize that some gut microbes persist over multiple generations and are adapted to varying degrees to their human hosts and families, making them potentially important members of the human gut. Bacterial strains can persist in the human host for years, with maternally-transferred strains known to persist longer in infants than environmentally acquired ones. It is conceivable that a given strain can colonize a host for several vertical generations, as already shown for Bifidobacterium using cultured isolates. Yet investigators currently lack knowledge of microbial persistence over multiple generations, and the proposed PEARL-AGE cohort is the first study investigating multi-generation persistence of gut bacteria (to our best knowledge).

The PEARL-AGE project will investigate microbial transfer and the evolution of microbes in family members from different generations. Investigators will recruit siblings, fathers/guardians, grandparents, and great-grandparents to fully capture vertical (between generations) and horizontal (same generation) microbial transmission across multiple generations, as well as tracking parallel microbial evolution in multiple family members. This will substantially increase our understanding of microbial transmission, long-term microbial persistence through generations and between cohabiting family members and siblings.

ELIGIBILITY:
Inclusion Criteria:

* The following relations of the PEARL mother/baby are eligible for inclusion:

  * Husband/partner of a PEARL mother, their biological parents and grandparents.
  * PEARL mother's biological parents and grandparents (great-grandparents to the PEARL baby).
  * Co-habiting non-biological fathers of the baby such as stepfathers and partners of the PEARL mother, their parents and grandparents.
  * A biological sibling of the PEARL baby or a step-sibling who is currently co-habiting with the PEARL baby.
* Adult participants must be able to consent for themselves and able to understand the questionnaire.
* Child participants must have a parent and/or guardian to provide assent on their behalf.
* Must be living in England.
* Must be willing to accommodate a small cool box to store and transport the biological samples until they are collected, if not having immediate access to the PEARL study freezer.
* Vulnerable participants such as participants with mild cognitive impairment may be included as long as they have full support from their family members.

Exclusion Criteria:

* Not related/affiliated to a mother currently participating in the PEARL study, or the cohabiting partner, or father of the PEARL infant. If a PEARL participant has withdrawn from the PEARL study or is no longer participating, investigators will not approach the PEARL participant for recruitment of their family members.
* Step-fathers or long-term partners that have been cohabiting with the PEARL mother for less than three months.
* Those currently in prison.
* Those who are unable to provide written informed consent.
* Living with or related to a member of the Research Study team.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Investigators are recruiting the family members of PEARL (ClinicalTrials.gov ID: NCT03916874) study participants, a longitudinal study to understand how gut microbes contribute to maintaining health during pregnancy and early life already underway at QIB (Quadram Institute Bioscience). Investigators will extend this cohort, by recruiting family members of the PEARL mother to form the PEARL-AGE cohort, extending it from two generations to four generations.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Characterizing microbial transfers in multigenerational families and subsequent stability of microbial colonization. | 2026
  High-resolution metagenomics of strains tracked over time in individuals and families, relative to collected metadata (family closeness, medical history, etc) Associating microbiome stability to human genetic loci.

SECONDARY OUTCOMES:
Characterizing gut microbial evolution and adaptation in human host families. | 2026
  Comparative genomics of metagenome assembled genomes (MAGs) per individual. Identifying newly introduced mutations in microbial genomes. Observing parallel evolution (e.g., loss or gain of the same genes in bacteria).
  Associating human genotypes to microbial adaptation.

OTHER OUTCOMES:
Describing the prokaryotic and eukaryotic genome-level diversity within the human gut | 2024
  Newly developed DNA extraction protocols for enrichment of specific microbial clades.
Identify predictors of within-family gut microbe transfer rates | 2026
  Correlation coefficient of collected metadata (questionnaire derived) to observed shared microbes Correlate parallel colonization's of sibling to family questionnaire metadata (e.g. distances, closeness, habits, ..) Correlate genetic factors (immune system, etc) to microbial sharing/colonization rates

CONTACTS AND LOCATIONS:
Overall Officials: Falk Hildebrand, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Biosciences, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided